CLINICAL TRIAL: NCT05360212
Title: Anatomy-based Fitting in Unexperienced Cochlear Implant Users. Programación Basada en la anatomía en Usuarios Nuevos de Implante Coclear.
Brief Title: Anatomy-based Fitting in Cochear Implant Users
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz (Other)
Collaborators: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Principal Investigator, Luis Lassaletta, Doctor, Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PI-6128
Record Dates: First submitted 2022-04-23; First posted 2022-05-04 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-02

CONDITIONS: Cochlear Implant; Outcomes; Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Standard fitting (Placebo Comparator): The first group is fitted using the standard frequency-band distribution as implemented in MAESTRO 9
  Interventions: Procedure: Standard Fitting
- Anatomy-based fitting (Experimental): In the second group of users, an anatomy-based frequency distribution is used as per anatomy-based fitting in MAESTRO 9
  Interventions: Procedure: Anatomy-based fitting (ABF)
- Within-subject design: Standard fitting + ABF (Experimental): The third group constitutes the within-subject design. These subjects are both fitting using the standard frequency-band distribution and the anatomy-based frequency distribution in MAESTRO 9. So, subjects will have both study maps on their audio processor throughout the whole study. They will have to change weekly between both fittings: standard fitting and anatomy-based fitting.
  Interventions: Procedure: Standard fitting+ ABF

INTERVENTIONS:
Procedure: Anatomy-based fitting (ABF) — MAESTRO 9 can display the tonotopic frequency of each individual electrode channel imported from OTOPLAN to further support fitting based on these measures. The audiologist can set a frequency-band distribution that is more closely aligned to the tonotopic frequency distribution as imported from OTOPLAN.
  Arms: Anatomy-based fitting
Procedure: Standard Fitting — These group is fitted using the standard frequency-band distribution as implemented in MAESTRO 9.
  Arms: Standard fitting
Procedure: Standard fitting+ ABF — Patients of this group are both fitting using the standard frequency-band distribution and the anatomy-based frequency distribution in MAESTRO 9. So, subjects will have both study maps on their audio processor throughout the whole study. They will have to change weekly between both fittings: standard fitting and anatomy-based fitting. Here, the performance with anatomy-based fitting is assessed by comparing performance with standard fitting and anatomy-based fitting.
  Arms: Within-subject design: Standard fitting + ABF

SUMMARY:
In this study, the performance with the CI is investigated over time in three groups of freshly implanted CI users. Both the standard frequency-band distribution and anatomy-based fitting will be used to compare outcomes.

DETAILED DESCRIPTION:
In this study, the performance with the CI is investigated over time in three groups of freshly implanted CI users. The first group is fitted using the standard frequency-band distribution as implemented in MAESTRO 9. In the second group of users, an anatomy-based frequency distribution is used as per anatomy-based fitting in MAESTRO 9. The performance with anatomy-based fitting is assessed by comparing performance with the CI in these two groups over time.

The third group constitutes the within-subject design. These subjects are both fitting using the standard frequency-band distribution and the anatomy-based frequency distribution in MAESTRO 9. So, subjects will have both study maps on their audio processor throughout the whole study. They will have to change weekly between both fittings: standard fitting and anatomy-based fitting. Here, the performance with anatomy-based fitting is assessed by comparing performance with standard fitting and anatomy-based fitting.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Post-lingual onset of severe to profound sensory-neural hearing loss in the implanted ear(s)
* Post-OP CT scan of the CI electrode available
* Subject implanted with MED-EL cochlear implant(s)
* Subjects received a Flex28 or FlexSoft electrode
* Subject planned to receive a SONNET 2 /RONDO3 audio processor on the newly implanted side
* Audio processor not yet activated on the newly implanted side
* The most apical active electrode contact has to be inserted at least 450°
* Minimum of 10 active channels can be activated
* Fluent in Spanish
* Signed and dated ICF before the start of any study-specific procedure

Specific inclusion criteria for the possible study groups • Bilateral CI users: Bilateral CI implantation SONNET 2/RONDO3 audio processor on the first ear implanted

* 40% speech recognition a monosyllabic word Test in quiet at 65 dB SPL (last time tested) on the already implanted side
* 40% speech recognition in a sentence test in noise (10 dB SNR) on the already implanted side First activation of the already implanted side between 3 and 12 months prior to study inclusion

  • Unilateral CI users: Unilateral CI implantation CI user with contralateral hearing ≥ 60 dB (PTA measured at 500, 1000, 2000, and 4000 Hz)

  • SSD CI users: Unilateral CI implantation CI user with contralateral hearing ≤30 dB (PTA measured at 500, 1000, 2000, and 4000 Hz) Interaural threshold gap ≥40 dB

  • Bimodal CI users: Unilateral CI implantation Contralateral ear adequately fitted with a hearing aid CI user with contralateral hearing ≥30 dB (PTA measured at 500, 1000, 2000, and 4000 Hz) CI user with contralateral hearing ≤55 dB (PTA measured at 500, 1000, 2000, and 4000 Hz) Interaural threshold gap ≥15 dB

Exclusion Criteria:

* Lack of compliance with any inclusion criteria
* EAS user (user of an EAS audio processor)
* Implanted with C40+, C40X and C40C
* Implanted with an ABI or Split electrode array
* Known allergic reactions to components of the investigational medical device
* Anything that, in the opinion of the Investigator, would place the subject at increased risk or preclude the subject's full compliance with or completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Result from the speech test in noise (S0N0) | Month 6
  Speech perception evaluation with CI-only (MATRIX) with signal and noise in the same channel
Results from speech tests in noise with spatially separated loudspeakers | Month 6
  Speech perception evaluation with CI-only (MATRIX) with signal and noise in different channels
Result from the speech test in quiet (S0) | Month 6
  Speech perception evaluation with CI-only (disyllables)

SECONDARY OUTCOMES:
Results of quality of sound | Month 6
  Subjective results through Hearing Implant Sound Quality Index 19. Scores range 19-133 points. Higher scores mean a better outcome.
Results of quality of life in challenging situations | Month 6
  Subjective results through Listening effort questionnaire. Scores range 21-93 points. Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Lassaletta, PhD, Principal Investigator — Fundacion para la Investigacion Biomedica del Hospital Universitario la Paz
Locations (1):
- Hospital Universitario de La Paz, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No